CLINICAL TRIAL: NCT06443164
Title: Efficacy of a Single-session Treatment for Reducing Chronic Pain Prior to Gender-affirming Surgery
Brief Title: Efficacy of a Chronic Pain Treatment Prior to Gender-affirming Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jenna Stapleton, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00026520
Record Dates: First submitted 2024-03-29; First posted 2024-06-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pain Catastrophizing; Pain, Chronic; Gender Identity
Keywords: Chronic Pain; Gender Diversity; Gender Affirming Surgery
MeSH Terms: conditions — Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Interventional Group Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Management Class (Experimental): Pain Management Class Prior to Gender Affirming Surgery
  Interventions: Behavioral: Empowered Relief
- SOC - No Class (Active Comparator): SOC for Gender Affirming Surgery
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Empowered Relief — Pain Management Course that has been used to treat pain in patients with different pain conditions.
  Arms: Pain Management Class
Other: Standard of Care — Gender Affirming surgery without any attention to pain conditions prior to surgery.
  Arms: SOC - No Class

SUMMARY:
The primary objective of this study is to examine a single-session, 2-hour group intervention provided to a population of transgender or gender-diverse patients with chronic pain prior to gender-affirming surgery, to determine if participants who receive the intervention have less pain-related distress compared to participants randomly assigned to the control group.

DETAILED DESCRIPTION:
The primary objective of this study is to examine a single-session, 2-hour group intervention provided to a population of transgender and gender-diverse patients with chronic pain prior to gender-affirming surgery, to determine if participants who receive the intervention have less pain-related distress compared to participants randomly assigned to the control group. This study will help extend the research literature on chronic pain experienced by transgender patients, and specifically will examine if a brief, group intervention is effective for reducing pain catastrophizing and pain distress prior to surgery.

Safety and effectiveness of the Empowered Relief intervention used in this study has been demonstrated in multiple clinical trials, but has not been studied yet with this particular population. The Empowered relief intervention was created by Beth Darnall © Stanford University.

The hypothesis of this research study is that transgender patients with chronic pain who receive the group intervention, prior to having a gender-affirming surgery, will have lower scores on the pain catastrophizing scale after completing the intervention compared to participants in the control group:

Hypothesis: µ1 <(<=) µ2. The primary endpoint of this study is to test if the mean change in the score on the Pain Catastrophizing Scale is different between the treatment and the control group. The secondary endpoint, is to examine if pain severity scores decreased. An exploratory endpoint, after data collection and analysis is complete, is to run a focus group with participants who received the intervention to learn more about their experience to inform future treatment and research. Safety endpoints are that participants will receive informed consent, which will include learning they may discontinue participation in the study at any time, as well as procedures for maintaining confidentiality of identifying information. Each person screened will already be referred to the Transgender Health Program by a primary care provider and/or mental health provider. If screening indicates that a person has severe depression or regular thoughts involving suicidal content, then that person will not be included in the study but instead will be offered resources and highly recommended to contact their referring provider for additional support.

ELIGIBILITY:
Inclusion Criteria:

1. affiliated with the OHSU Transgender Health Program and have completed their initial consultation for gender-affirming surgery,
2. who have chronic pain (defined as > 3 months of pain),
3. who rate their average level of pain intensity as at least a 4 or higher (on 0-10 pain scale)
4. who have fluency in English. Empowered Relief may only be delivered by a certified instructor, and for this research study the instructor is only able to offer the curriculum in English.

Exclusion Criteria:

1. have had a pain-focused behavioral therapy in the past year, or
2. have severe depression and/or moderate or higher risk of suicidality based on the person's score on the PHQ-9 greater than 20.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Anyone who identifies as gender diverse or transgender and seeking gender affirming surgical care.
Enrollment: 78 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing | Participants will be assessed as part of a cohort for up to 7 months. There will be a total of three cohorts.
  This measure is a 13-item self-assessment instrument of pain-related negative thoughts, and measures constructs of rumination, magnification and helplessness. It is the primary outcome measure of this research study. Each item is measured on a 5-point Likert scale, with endpoints 0 (not at all) to 4 (all the time) and possible scores ranging from 0-52. In a clinical setting, such as a pain clinic providing treatments for chronic pain, a score on this measure of "10" or higher indicates a person could benefit from treatment; however, the published cut-off scores are higher and as follows: a Total Score of 20 is considered in the average range (50th percentile), and a Total Score of >= 30 is above average (75th percentile). This measure is shown to have excellent internal consistency (coefficient alphas: total PCS = .87, rumination = .87, magnification = .66, and helplessness = .78.

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU Comprehensive Pain Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
If information is shared in the future outside OHSU it will be deidentified and shared as a data set.

REFERENCES:
- [Derived] Stapleton JW, Bohacek SH, Marsiglio M, Kachmarik JE, Carson JW. Efficacy and feasibility of a telehealth intervention (Empowered Relief) for reducing pain-related discouraging thoughts and emotions for gender-diverse adults prior to surgery: protocol for a randomized controlled trial. BMC Surg. 2025 Dec 17. doi: 10.1186/s12893-025-03423-5. Online ahead of print. PMID 41402818